CLINICAL TRIAL: NCT05939882
Title: A Double-blind, Randomized Controlled Study of Low Concentration Atropine in the Prevention of Myopia in Pre-myopia Children.
Brief Title: Low Concentration Atropine in the Prevention of Myopia in Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: jafakfakfa
Record Dates: First submitted 2023-06-23; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.01% atropine (Experimental): 0.01% atropine eye drop
  Interventions: Drug: low concentration atropine (0.01%)
- 0.02% atropine (Experimental): 0.02% atropine eye drop
  Interventions: Drug: low concentration atropine (0.02%)
- 0.04% atropine (Experimental): 0.04% atropine eye drop
  Interventions: Drug: low concentration atropine (0.04%)
- placebo (Placebo Comparator): placebo eye drop
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: low concentration atropine (0.01%) — low concentration atropine (0.01%)
  Arms: 0.01% atropine
Drug: low concentration atropine (0.02%) — low concentration atropine (0.02%)
  Arms: 0.02% atropine
Drug: low concentration atropine (0.04%) — low concentration atropine (0.04%)
  Arms: 0.04% atropine
Drug: Placebo — Placebo eye drop
  Arms: placebo

SUMMARY:
This double-blind, randomized controlled clinical study is to evaluate the effectiveness and safety of low concentration atropine in preventing myopia in pre-myopia children, and to explore whether there is a dose effect relationship between different concentrations of atropine in preventing myopia.

DETAILED DESCRIPTION:
The main questions this double-blind, randomized controlled clinical study aims to answer are:

1. To evaluate the effect of low concentration atropine on the incidence of myopia in pre myopia children.
2. To evaluate the effectiveness of low concentration atropine in controlling refractive and axial progression.

Patients are randomly divided into three treatment groups with different atropine concentrations(0.01%, 0.02%, 0.04%) and one control group with atropine dissolvant. Patients are required to use the eye drops every night for one year and record after daily usage.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the screening stage is 6-9 years, both sexes;
2. One eye met the diagnosis of pre-myopia, the spherical equivalent was between -0.50D and +0.75D, the astigmatism was ≥-1.50D, and the best corrected far vision was at least 1.0;
3. At least one of parents suffers from myopia (SE of at least one eye <=-3.00D);
4. Parents have signed informed consent and agree to participate in screening and follow-up.

Exclusion Criteria:

1. Parents disagree to sign the informed consent;
2. Presence of strabismus, amblyopia, or other ocular abnormalities, or have a history of eye surgery;
3. Presence of other eye or systemic diseases;
4. Allergies to low concentration atropine or sulfuric acid drugs;
5. Histories of using other preventive measures, such as using red light within 6 months or atropine within 1 month;
6. Presence of other situations that the researchers think is not appropriate for patients to be included in the project.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 428 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Cumulative Incidence of Myopia | 1 year
  Effectiveness Evaluation

SECONDARY OUTCOMES:
Changes in SE (after cycloplegia) | 1 year
  Effectiveness Evaluation
Changes in AL | 1 year
  Effectiveness Evaluation
Changes in visual acuity | 1 year
  Effectiveness Evaluation
Changes in Choroidal Thickness | 1 year
  Effectiveness Evaluation

OTHER OUTCOMES:
Changes in Photophobia Incidence Rate | 1 year
  Safety Evaluation
Changes in Blurred Vision Incidence Rate | 1 year
  Safety Evaluation
change in amplitude of accommodation | 1 year
  Safety Evaluation
change in pupil size | 1 year
  Safety Evaluation
change in ocular surface health | 1 year
  Safety Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: He Xiangui, Study Director — Shanghai Eye Disease Prevention and Treatment Center
Locations (1):
- Xiangui He, Shanghai, Shanghai Municipality, China